CLINICAL TRIAL: NCT06570382
Title: Evaluating Taste and Health Messaging in Short Nutrition Education Videos on Increasing Herb and Spice Use to Improve Diet Quality
Brief Title: Evaluating Taste and Health Messaging in Short Nutrition Education Videos to Improve Diet Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Travis Masterson, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00025218
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taste video participants (n=500) (Active Comparator): Participants in this arm will only watch taste focused messaging videos
  Interventions: Other: Videos: Taste messaging focused
- Health video participants (n=500) (Active Comparator): Participants in this arm will only watch health focused messaging videos.
  Interventions: Other: Videos: Health messaging focused

INTERVENTIONS:
Other: Videos: Taste messaging focused — Participants in this intervention will watch the taste focused videos.
  Arms: Taste video participants (n=500)
Other: Videos: Health messaging focused — Participants in this intervention will watch the health focused videos.
  Arms: Health video participants (n=500)

SUMMARY:
The purpose of this study is to develop and evaluate the effectiveness of taste vs. health messaging using nutrition education videos. The nutrition education videos teach Americans the benefits of using herbs and spices to increase diet quality. The investigators aim to test the effectiveness of 10 short videos (5 taste-based messaging and 5 health-based messaging) that translate previous findings of how spices can improve diet quality. These objectives will be pursued via the following hypothesis:

Hypothesis 1: Are taste messaging videos more effective in improving consumer interest, knowledge, and confidence in using herbs and spices compared to health messaging focused videos? Hypothesis 2: Will consumers rate the taste messaging videos higher for liking, engagement, and acceptability of herbs and spices compared to health messaging focused videos?

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two groups: the first group (n=500) will receive the taste messaging focused videos emphasizing taste and flavor, while the second group (n=500) will receive the health messaging focused videos emphasizing the importance of using herbs to improve health. Randomization will occur through REDCap and the randomization feature will be embedded in the survey. Both groups will have access to similar educational content but the focus of the messaging will differ according to the taste or health focused arm. The participants will also complete screening questions first, and if eligible, an online consent form, demographics questionnaire, pre implementation questionnaire via REDCap, data on the participants interest, knowledge and confidence in using spices and herbs before watching the video and then watch 5 videos of either the taste or health focused messaging video (dependent on randomization). Once completed, participants will then complete a post implementation questionnaire, and a post-intervention REDCap survey that will ask about their interest, knowledge and intent in using spices and herbs as well as their feedback on the effectiveness of the videos. The investigators will use the pre and post intervention surveys for analysis. All participants will complete the survey questions online using their own device. The survey will also include more detailed participant information and gather feedback on the implementation of recipes in their own kitchens.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-75 years of age
* Reside in the United States
* Fluent in English
* Have access to internet, a video viewing device (computer, phone, tablet, etc.), and a grocery store
* Able to cook at home at least 2x/week or more

Exclusion Criteria:

* Outside of the 18-75 year age range
* Resides outside the United States
* Are not fluent in English
* Does not have access to internet or video viewing device (computer, phone, tablet, etc.), or a grocery store
* Unable to cook at home at least 2x/week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
Ratings for interest, knowledge, confidence variables in using herbs and spices in cooking from before to after exposure to nutrition education videos using Likert scales from 0-5 with 0 being strongly disagree to 5 being strongly agree. | Within 5 minutes of watching the nutrition education videos
  Participants will provide feedback on the taste and health-based messaging videos which will be used to create more effective messaging in the subsequent video development.

SECONDARY OUTCOMES:
Ratings for liking, engagement, and acceptability of using herbs and spices in cooking from before to after exposure to nutrition education videos using Likert scales from 0-5 with 0 being strongly disagree to 5 being strongly agree. | Within 5 minutes of watching the nutrition education videos
  Participants will provide feedback on the taste and health-based messaging videos which will be used to create more effective messaging in the subsequent video development.

CONTACTS AND LOCATIONS:
Locations (1):
- Dynata Online Market Research Agency, Shelton, Connecticut, United States